CLINICAL TRIAL: NCT05600179
Title: Evaluation of Changes in Epivascular Glia Before and After Intravitreal Dexamethasone Implant : an OCT Pilot Study
Brief Title: OCTA in Epivascular Glia After Dex Implant
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, professor, Federico II University
Other Study IDs: 0110/2022
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with diabetic macular edema
  Interventions: Drug: Dexamethasone intravitreal implant
- healthy patients

INTERVENTIONS:
Drug: Dexamethasone intravitreal implant — Dexamethasone intravitreal implant
  Groups: patients with diabetic macular edema

SUMMARY:
The aim of this prospective study was for the first time, to analyze specific morphologic features in diabetic eyes with macular oedema, such as changes of the foveal avascular zone and the presence of epivascular glia, and see how they would change after dexamethasone intravitreal implant

ELIGIBILITY:
Inclusion Criteria:

* diabetic retinopathy complicated by macular edema

Exclusion Criteria:

* congenital eye disorders,
* previous diagnosis of other ocular diseases
* history of vitreous hemorrhage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participans were older than 18 years with diagnosis of inflammatory diabetic macular edema glaucoma..
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in epivascular glia after Dexamethasone implant in patients with diabetic retinopathy and inflammatory macular edema | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples "Federico II", Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes